CLINICAL TRIAL: NCT05795855
Title: An Adaptive Prenatal Intervention to Increase Childhood Vaccinations
Acronym: ADEPT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is suspended pending a protocol amendment.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lavanya Vasudevan, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005432; STUDY00005431 (Other: Emory University); U01IP001149 (NIH); STUDY00005457 (Other: Emory University)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Vaccination Refusal
Keywords: Vaccine hesitancy
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADEPT (Experimental): Individuals receiving prenatal care at a practice that was randomized to deliver the ADEPT intervention.
  Interventions: Behavioral: ADEPT
- Standard of Care (No Intervention): Individuals receiving prenatal care at a practice that was randomized to deliver the standard of care.

INTERVENTIONS:
Behavioral: ADEPT — Prenatal providers will participate in trainings that will lay the foundation for an effective vaccination recommendation. After the completion of training, prenatal care providers will begin making recommendations promoting the importance of maternal and childhood vaccinations to pregnant individuals, as part of routine prenatal care. The core component of ADEPT is prenatal provider training to enable a vaccination recommendation, encouraging pregnant individuals to receive vaccines during pregnancy and for their child after birth. Pregnant individuals who remain vaccine hesitant despite the provider recommendation, will be eligible to receive the adaptive components of ADEPT in the form of evidence-based educational materials on vaccinations and phone consultations with a vaccine navigator to discuss residual concerns.
  Arms: ADEPT

SUMMARY:
This study will test whether proactively connecting expectant parents with factual vaccination information during pregnancy can build confidence in vaccinations and lead to timely vaccinations during pregnancy and once their child is born.

DETAILED DESCRIPTION:
In the United States (US), parents' decision to delay or refuse vaccines for their children has resulted in pockets of under-vaccination as well as recurring outbreaks of vaccine-preventable diseases. To increase childhood vaccinations and stem recurring outbreaks, there is a need for effective interventions that build parents' confidence in vaccines and reduce their vaccine hesitancy. The first recommended routine vaccination for children is due at birth. Yet, many parents lack timely or evidence-based information on childhood vaccinations prior to their child's birth. Hence, the researchers of this study propose to evaluate ADEPT - an adaptive intervention that is implemented in prenatal care settings to proactively connect expectant parents with evidence-based information on vaccines recommended during pregnancy and for children after birth. The core component of ADEPT includes prenatal provider trainings and a recommendation to pregnant individuals encouraging vaccinations during pregnancy and for children after birth. Those pregnant individuals who remain vaccine-hesitant despite the provider recommendation will receive adaptive intervention components, which include evidence-based educational materials on vaccinations and phone consultations with a vaccine navigator to discuss any residual concerns.

In the proposed study, ADEPT will be implemented and evaluated in diverse prenatal care practices in North Carolina. Study prenatal care practices will be randomized to the ADEPT intervention or standard of care to pregnant individuals. Individuals receiving prenatal care at a clinic implementing ADEPT will be screened for vaccination intention following the provider recommendation. Vaccine-hesitant pregnant individuals will be offered enrollment into a nested sub-study designed to assess the implementation of the ADEPT intervention. After the pregnant individuals in the intervention and control arms give birth, the researchers will assess their children's vaccination outcomes at birth, 2, 4, 6, and 12 months using data from the North Carolina Immunization Registry (NCIR). The primary study outcome is the difference in timely childhood vaccination at 2 months between the intervention and control arms. In addition, maternal vaccination data will be collected from NCIR for vaccines during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous individuals (no prior live birth)
* Singleton pregnancy (excludes twins, triplets, etc.)
* No known fetal congenital malformations or genetic abnormalities
* Not at known risk for preterm birth
* In late second trimester during study recruitment period
* Receive prenatal care at one of the study practices

Inclusion Criteria for Nested Sub-Study:

* Eligible to receive adaptive components of ADEPT (vaccine-hesitant after provider recommendation)
* At least 18 years of age
* Provide informed consent
* Agree to participate in surveys and in-depth interview
* Agree for child's vaccination outcomes to be extracted from the North Carolina Immunization Registry (NCIR)
* Plan to stay in North Carolina for at least 3 months after delivery

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children receiving timely vaccinations | 2 months post birth
  The proportion of children who receive vaccinations per the Advisory Committee on Immunization Practices (ACIP) recommended schedule at 2 months-post birth, by study arm.

SECONDARY OUTCOMES:
Change in Vaccine Hesitancy | 28-32 weeks gestation (after receiving the core ADEPT intervention), following completion of the adaptive portion of ADEPT (prior to birth, typically 40 weeks gestation)
  In the intervention arm only, vaccine hesitancy will be examined among pregnant individuals in the intervention prenatal practices. When asked about vaccination intention, lack of intention to get vaccinations during pregnancy or for their child after birth will determine if they will receive the adaptive portion of ADEPT. The question will be asked again following completion of the ADEPT adaptive components.

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Vasudevan, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Duke Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets related to the primary outcome will be made available after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Dataset will be posted after publication of manuscript describing the primary outcome, with no end date.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Proposals should be directed to lavanya.vasudevan@emory.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Derived] Vasudevan L, Porter RM, Campos I, Turner EL, Stinnett SS, Zullig LL, Walter EB, Swamy GK, Bednarczyk RA, Orenstein WA, Gray B. An ADaptivE PrenaTal (ADEPT) intervention to increase childhood vaccinations: Protocol for a cluster randomized trial and nested mixed methods evaluation. PLoS One. 2024 Nov 21;19(11):e0313742. doi: 10.1371/journal.pone.0313742. eCollection 2024. PMID 39570957